CLINICAL TRIAL: NCT00351221
Title: A Phase 2, Open-Label, Multicenter, Clinical Trial to Evaluate the Pharmacokinetics, Safety and Efficacy of Recombinant Human Insulin-Like Growth Factor-1/Recombinant Human Insulin-Like Growth Factor Binding Protein-3 in Children With Growth Failure Due to Noonan Syndrome
Brief Title: Research Study Using Recombinant Human Insulin-Like Growth Factor-1/Recombinant Human Insulin-Like Growth Factor Binding Protein-3 for Children With Noonan Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to a patent legal settlement
Sponsor: Insmed Incorporated (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INMS-110-801
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2007-03-30 (Estimated); Status verified 2007-02

CONDITIONS: Noonan Syndrome
MeSH Terms: conditions — Noonan Syndrome

INTERVENTIONS:
Drug: rhIGF-1/rhIGFBP-3

SUMMARY:
The trial will investigate the treatment of growth failure in children with Noonan syndrome. Abnormalities in the growth hormone (GH) - insulin-like growth factor-I (IGF-I) axis resulting in low IGF-I levels have been suggested as a possible cause of short stature seen in Noonan syndrome children. Administration of our investigational product is intended to bypass the abnormalities in the GH-IGF axis, and hopefully improve body growth.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of Noonan syndrome
2. Height less than the 3rd percentile for age and sex (height SDS < -1.88)
3. Basal IGF-I less than the mean for age and sex (IGF-I SDS < 0)
4. Chronological age greater than 2 years
5. Bone age ≤ 11 years for boys, and ≤ 10 years for girls
6. Pre-pubertal
7. Documented pre-treatment height velocity less than the mean for age and sex

Exclusion Criteria:

1. Clinically significant diseases
2. Chronic illnesses
3. Prior treatment with rhIGF-1

Ages: 2 Years to 16 Years | Sex: All
Age Groups: Child
Enrollment: 24

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Attie, MD, Study Director — Insmed, Inc.
Locations (2):
- United States (2):
  - Schneider Children's Hospital, New Hyde Park, New York
  - Columbus Children's Hospital, Columbus, Ohio